CLINICAL TRIAL: NCT04294745
Title: Effectiveness of Buccal Infiltration and Inferior Alveolar Nerve Block With Articaine for Extraction of Mandibular Teeth- A Randomized Clinical Trial
Brief Title: Comparing Buccal Infiltration and Inferior Alveolar Nerve Block for Extraction of Mandibular Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Abdul Kalam Azad, Assistant Professor, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMMC/FOD/AR/B7/E C-2019 (04)
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Buccal Infiltration Inferior Alveolar Nerve Block Articaine
Keywords: Buccal infiltration inferior alveolar nerve block Articaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Buccal infiltration of 4% Articaine
  Interventions: Procedure: Buccal infiltration
- Group B (Active Comparator): Inferior alveolar nerve block of 4% Articaine
  Interventions: Procedure: Inferior alveolar nerve block

INTERVENTIONS:
Procedure: Buccal infiltration — Injection of local anaesthetic parallel to the Long axis of the tooth in the depth of buccal sulcus
  Arms: Group A
Procedure: Inferior alveolar nerve block — Standard technique of mandibular nerve block
  Arms: Group B

SUMMARY:
This study compares the effectiveness of two techniques of local anesthesia in the extraction of mandibular teeth. One group received inferior alveolar nerve block and the other group received buccal infiltration of 4% Articaine

DETAILED DESCRIPTION:
Inferior alveolar nerve block is the commonly used local anesthetic injection technique for extraction of mandibular teeth. Buccal infiltration technique alone is considered to be ineffective in treating mandibular teeth due to the thickness of buccal cortical plate. However, buccal infiltration, if provided with an agent with higher penetration capability, may be used instead of Inferior alveolar nerve block. Articaine, due to its thiophene ring, has higher liposolubility and bony diffusion than any other agent.

This study compares the effectiveness of inferior alveolar nerve block and buccal infiltration using 4% Articaine in the extraction of mandibular teeth

ELIGIBILITY:
Inclusion Criteria:

* Mandibular teeth
* grossly decayed teeth
* root stumps
* therapeutic extractions
* American society of anesthesiologist classification I & II patients

Exclusion Criteria:

* patients allergic to local anesthesia
* infected teeth
* grade 2 and grade 3 mobile teeth
* patients already taking medications which influences the anaesthetic assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Pain during injection using a visual analogue scale measuring 10 cm with 0 depicting no pain and 10 depicting severe pain | During injection
  VAS scale is a validated scale measuring pain with possible score range from 0 (no pain) to 10 (severe pain).
Pain during extraction using a visual analogue scale measuring 10 cm with 0 depicting no pain and 10 depicting severe pain | During extraction
  VAS scale is a validated scale measuring pain with possible score range from 0 (no pain) to 10 (severe pain).
Requirement of rescue injection | During extraction
  whether a recue injection was given or not

CONTACTS AND LOCATIONS:
Overall Officials: Abdul R Ismail, Study Director — Melaka Manipal Medical College
Locations (1):
- Melaka Manipal Medical College, Malacca, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 1 month
Access Criteria: Study protocol will be provided only if requested through a proper channel , dean of the college, with proper justification.